CLINICAL TRIAL: NCT04202614
Title: Prognostic Role of Positron Emission Tomography and Computed Tomography Parameters in Stage I Lung Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Carretta Angelo, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PET-TC Adenocarcinoma
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Stage I Pulmonary Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical and derived data from the preoperative computed axial tomography (CT) and Positron Emission Tomography (PET) of patients with pathological stage I pulmonary adenocarcinoma will be analyzed retrospectively, classified according to the current pathological classification IASLC / ATS / ERS of pulmonary adenocarcinoma, subjected to surgical treatment in our Operating Unit between August 2006 and July 2011. A follow-up will be performed on the patients enrolled in the study up to the date of death, and in any case no later than October 31, 2019

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from pulmonary adenocarcinoma in stage I underwent CT, PET and surgical treatment with radical intent, at San Raffale Hospital (thoracic surgery) between August 2006 and July 2011

Exclusion Criteria:

* primary pulmonary neoplasms other than adenocarcinoma; locally advanced or metastatic disease stage; non-radical resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from pulmonary adenocarcinoma in stage I
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Stratification of stage I adenocarcinoma patients, using clinical data derived from preoperative CT and PET | 12 months
  classify patients with pulmonary adenocarcinoma in stage I (retrospective cases) based on the current pathological classification IASLC / ATS / ERS of pulmonary adenocarcinoma using clinical data and derived from preoperative CT and PET

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khullar OV, Liu Y, Gillespie T, Higgins KA, Ramalingam S, Lipscomb J, Fernandez FG. Survival After Sublobar Resection versus Lobectomy for Clinical Stage IA Lung Cancer: An Analysis from the National Cancer Data Base. J Thorac Oncol. 2015 Nov;10(11):1625-33. doi: 10.1097/JTO.0000000000000664. PMID 26352534
- [Result] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008
- [Result] Tsutani Y, Miyata Y, Nakayama H, Okumura S, Adachi S, Yoshimura M, Okada M. Appropriate sublobar resection choice for ground glass opacity-dominant clinical stage IA lung adenocarcinoma: wedge resection or segmentectomy. Chest. 2014 Jan;145(1):66-71. doi: 10.1378/chest.13-1094. PMID 24551879